CLINICAL TRIAL: NCT07000513
Title: Innovative Tools to Expand HIV Self-Testing and Long-Acting Injectables for HIV Treatment and Prevention Among Commercial Minibus Drivers (I-TEST LAIs)
Brief Title: HIV Self-Testing and Long-Acting Injectables for HIV Treatment and Prevention Among Commercial Minibus Drivers (I-TEST LAIs) in Nigeria
Acronym: ITEST-LAI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: The George Washington University Milken Institute School of Public Health (GWU) (Unknown)
Responsible Party: Principal Investigator, Donaldson Conserve, Multiple Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR245734; 1R01AI186786-01 (NIH)
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: HIV; PrEP; Long-acting Injectables; Nigeria; Minibus drivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-TEST LAI Intervention: (Experimental): Participants enrolled in the intervention arm will receive instructions on HIVST and HIVST bundles from MPERFs at the motor parks after completing the baseline survey. Participants will receive HIVST bundles which will contain 3 HIVST kits with a mobile photo-verification application or USSD-Unstructured Supplementary Service Data for uploading their results and access to the nearest male-friendly health clinics. MPERFs will provide participants with instructions on how to use the photo verification application to report their results during each distribution period. During the HIVST bundle distribution and HIVST results reporting, MPERFs will also share information about the nearby male-friendly clinics and explain to the participants the need for visiting these clinics for confirmatory HIV testing. MPERFs will also provide information about the information about the benefits of LAI PrEP and LAI ART and offer to accompany participants to their appointments.
  Interventions: Behavioral: ITEST-LAI
- Standard of Care (No Intervention): Participants at motor parks randomized to the control group will receive flyers distributed at the motor parks from the study team member at baseline, and during the follow-up surveys with information about HIV testing, including HIVST, and information about the two male-friendly clinics nearby where they can get tested for HIV, collect HIVST kits, and initiate oral or LAI ART or PrEP. All clinic staff in the SoC arm will receive training on LAI ART and LAI PrEP and the clinics will be equipped with LAI ART and LAI PrEP as well as oral ART and oral PrEP for study participants. Participants will be reminded during follow-up surveys about these clinics and receive additional flyers with information about these clinics and the availability of HIVST and LAIs at these services. The MPERFs will only contact SoC participants for follow-up surveys and to collect their HIVST results if they visit the clinics to collect the HIVST kits.

INTERVENTIONS:
Behavioral: ITEST-LAI — The ITEST-LAI intervention includes male peer-led HIVST distribution and promotion, linkage to male-friendly clinics for confirmatory testing and follow-up care, peer support and technical assistance to address implementation challenges, and continuous monitoring and feedback for male peer educators and research facilitators (MPERFs).
  Arms: I-TEST LAI Intervention:

SUMMARY:
Long-acting injectable antiretroviral therapy (LAI ART) and Pre-Exposure Prophylaxis (LAI PrEP) have the potential to transform HIV treatment and prevention, especially in reaching individuals such as commercial minibus drivers who have minimal or no contact with traditional health facilities. The project proposes to use a culturally appropriate and community-engaged approach to promote the uptake of HIV self-testing, LAI-ART, and LAI-PrEP among commercial minibus drivers in Nigeria by engaging commercial minibus drivers as peer educators/research facilitators.

DETAILED DESCRIPTION:
Commercial minibus drivers constitute a large social network of highly mobile men who work long and demanding hours, are at increased risk for HIV, and have limited time to seek health services for HIV. In our preliminary work, our team found a high HIV seropositivity rate of 12.5% among 407 commercial minibus drivers in Nigeria, a prevalence that is nine times higher than the national HIV average. Despite the high willingness to test for HIV among the drivers, the mobile nature of their work poses substantial barriers for those living with HIV to initiate and adhere to antiretroviral therapy (ART) and for those who are HIV-negative and are at risk for HIV to obtain pre-exposure prophylaxis (PrEP). Therefore, innovative strategies such as HIV self-testing (HIVST), which allows individuals to test at home or in private, and long-actinginjectable ART (LAI ART) or LAI PrEP may work better to address the barriers that impede commercial drivers from accessing HIV testing, prevention, and treatment services. The investigators have recently evaluated a youth-friendly HIVST intervention combined with linkage to PrEP in Nigeria as part of an NIH-funded project called ITEST: Innovative Tools to Expand Youthfriendly HIV Self-Testing (UH3HD096929). The investigators propose to leverage our established research program in Nigeria in collaboration with the National Institute of Medical Research to implement a tailored ITEST intervention for commercial minibus drivers (ITEST LAIs), which will include male peer-led distribution of HIV self-testing kits combined with demand creation for both oral and LAI modalities of ART and PrEP. The multi-disciplinary research team proposes a hybrid type I effectiveness-implementation study to assess clinical and implementation determinants outcomes simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Male commercial minibus drivers who have worked as a driver for at least 6 months
2. 18 years old or older
3. Currently and planning on residing in one of the LGAs during the next 12 months
4. Owning a mobile phone

Exclusion Criteria:

1. Known HIV positivity
2. Not ability to provide informed consent3
3. No access to a cell phone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
ART or PrEP Initiation | Baseline and follow-up surveys at 6-,12-, 18-, and 24 months
  Use of patient records and self-report to determine initiation of HIV treatment or preventive medications.

SECONDARY OUTCOMES:
HIV Testing | Baseline and follow-up surveys at 6-,12-, 18-, and 24-months
  Use of patient records and self-report to determine HIV testing behavior (including use of HIVST and confirmatory testing in clinics).
ART Adherence | Baseline and follow-up surveys at 6-,12-, 18-, and 24-months
  Use of self-report and hair sample to measure medication adherence.
PrEP Adherence | Baseline and follow-up surveys at 6-,12-, 18-, and 24-months
  Use of hair samples and self-report to measure medication adherence.
Viral Load Supression | Baseline and follow-up surveys at 6-,12-, 18-, and 24-months
  Use of blood samples to measure viral load suppression among those who received an HIV diagnosis.
HIV Acquisition | Baseline and follow-up surveys at 6-,12-, 18-, and 24-months
  Use of blood samples, self-report, and patient records to measure seroconversion among study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Medical Research, Lagos, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared given the confidential nature of this study and terms under which participants agree to enroll.

REFERENCES:
- [Background] Majam M, Conserve DF, Zishiri V, Haile ZT, Tembo A, Phiri J, Hatzold K, Johnson CC, Venter F. Implementation of different HIV self-testing models with implications for HIV testing services during the COVID-19 pandemic: study protocol for secondary data analysis of the STAR Initiative in South Africa. BMJ Open. 2021 May 18;11(5):e048585. doi: 10.1136/bmjopen-2020-048585. PMID 34006558
- [Background] Iwelunmor J, Tucker JD, Obiezu-Umeh C, Gbaja-Biamila T, Oladele D, Nwaozuru U, Musa AZ, Airhihenbuwa CO, Muessig K, Rosenberg N, BeLue R, Xian H, Conserve DF, Ong JJ, Zhang L, Curley J, Nkengasong S, Mason S, Tang W, Bayus B, Ogedegbe G, Ezechi O. The 4 Youth by Youth (4YBY) pragmatic trial to enhance HIV self-testing uptake and sustainability: Study protocol in Nigeria. Contemp Clin Trials. 2022 Mar;114:106628. doi: 10.1016/j.cct.2021.106628. Epub 2021 Nov 17. PMID 34800699